CLINICAL TRIAL: NCT00224055
Title: A Randomized, Controlled, Open-label Study of the Safety and Efficacy of Ferrlecit® vs Oral Iron in Iron Deficient Patients With Chronic Kidney Disease
Brief Title: Effect of Ferrlecit® Versus Oral Iron on Iron Deficient Chronic Kidney Disease (CKD) Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Watson Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FER0202
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Results first posted 2012-03-29 (Estimated); Last update posted 2012-03-29 (Estimated); Status verified 2012-02

CONDITIONS: Anemia, Iron-Deficiency; Kidney Failure, Chronic
Keywords: Iron deficiency; Anemia; Chronic kidney disease; Sodium Ferric Gluconate; Anemia, Iron-Deficiency/drug therapy/etiology; Kidney Failure, Chronic/blood/complications/therapy
MeSH Terms: conditions — Anemia, Iron-Deficiency; Kidney Failure, Chronic; Iron Deficiencies; Anemia; Renal Insufficiency, Chronic; Renal Insufficiency; Bronchiolitis Obliterans Syndrome | interventions — ferric gluconate; Sucrose; Iron-Dextran Complex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IV iron (Experimental): Sodium ferric gluconate
  Interventions: Drug: Sodium Ferric Gluconate Complex in Sucrose Injection
- oral iron (Active Comparator): ferrous sulfate
  Interventions: Drug: Ferrous sulfate tablets

INTERVENTIONS:
Drug: Sodium Ferric Gluconate Complex in Sucrose Injection — Sodium Ferric Gluconate Complex in Sucrose Injection (Ferrlecit®), 250 mg IV weekly for 4 weeks
  Arms: IV iron
Drug: Ferrous sulfate tablets — ferrous sulfate, 325 mg oral, three times daily for 6 weeks
  Arms: oral iron

SUMMARY:
This study compares the effect of Ferrlecit® (a form of intravenous iron) to ferrous sulfate (a form of oral iron) in treating anemia and iron deficiency in chronic kidney disease patients who are not receiving erythropoietic agents (hormones that stimulate the bone marrow to make more red blood cells).

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe anemia
* Iron deficiency
* Moderate to severe chronic kidney disease

Exclusion Criteria:

* Receiving dialysis
* Known sensitivity to Ferrlecit® or any of its components
* Receiving therapy with erythropoietic agent
* Clinically unstable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2003-04; Primary Completion 2004-09 (Actual); Study Completion 2004-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Dahl, Pharm.D., Study Director — Watson Laboratories, Inc.
Locations (24):
- United States (23):
  - Tucson, Arizona
  - Los Angeles, California
  - Palo Alto, California
  - San Diego, California
  - Hines, Illinois
  - Indianapolis, Indiana
  - Shreveport, Louisiana
  - Baltimore, Maryland
  - Springfield, Massachusetts
  - Detroit, Michigan
  - St Louis, Missouri
  - Birmingham, New York
  - Mineola, New York
  - New York, New York
  - The Bronx, New York
  - Chapel Hill, North Carolina
  - Cleveland, Ohio
  - Philadelphia, Pennsylvania
  - Charlotte, South Carolina
  - Chattanooga, Tennessee
  - Memphis, Tennessee
  - Houston, Texas
  - Fairfax, Virginia
- San Juan, Puerto Rico

REFERENCES:
- [Result] Agarwal R, Rizkala AR, Bastani B, Kaskas MO, Leehey DJ, Besarab A. A randomized controlled trial of oral versus intravenous iron in chronic kidney disease. Am J Nephrol. 2006;26(5):445-54. doi: 10.1159/000096174. Epub 2006 Oct 11. PMID 17035697

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IV Iron | Oral Iron
Started | 44 | 45
Completed | 29 | 31
Not Completed | 15 | 14
Not completed — Adverse Event | 9 | 3
Not completed — Lost to Follow-up | 1 | 2
Not completed — Protocol Violation | 1 | 1
Not completed — Inclusion Violation | 3 | 6
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IV Iron | Oral Iron | Total
Number analyzed (Participants) | 44 | 45 | 89
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 19 | 48
  >=65 years | 15 | 26 | 41
Age Continuous [Mean (Standard Deviation); unit: years] | 66.3 (12.27) | 62.6 (14.86) | 64.4 (13.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 25 | 49
  Male | 20 | 20 | 40
Region of Enrollment [Number; unit: participants]
  United States | 43 | 44 | 87
  Puerto Rico | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemoglobin (Hgb)
Description: Change from baseline to 7 weeks after 4 consecutive weekly Ferrlecit 250 mg intravenious infusion and change from baseline to 4 weeks after 6 weeks oral ferrous sulfate 325 mg tablets t.i.d.
Time Frame: Baseline to 10 weeks
Population: Modified ITT with LOCF imputation
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | IV Iron | Oral Iron
Number analyzed (Participants) | 36 | 39
g/dL | 0.6 (0.94) | 0.2 (1.11)

2. Secondary Outcome: Change in Serum Ferritin
Description: as for outcome 1
Time Frame: Baseline to 10 weeks
Population: Modified ITT with LOCF imputation
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | IV Iron | Oral Iron
Number analyzed (Participants) | 36 | 39
ng/mL | 207.7 (207.02) | 22.6 (53.40)

ADVERSE EVENTS:
Arm/Group | IV Iron | Oral Iron
Serious Adverse Events (participants affected / at risk) | 4/44 | 4/45
Other Adverse Events (participants affected / at risk) | 22/44 | 21/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IV Iron (N=44) | Oral Iron (N=45)
Exacerbation Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Lower Exteremities Skin Abcess Lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
Worsening Chronic Kidney Disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Anaphylaxis (Immune system disorders) | 1 (1) | 0 (0)
Bilateral Pleural Iffusions (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute Renal Failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Admitted to Hospital for Renal Biopsy (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IV Iron (N=44) | Oral Iron (N=45)
Abdominal Enlargement (General disorders) | 0 | 3
Asthenia (General disorders) | 1 | 3
Infection (Infections and infestations) | 2 | 3
Abdominal Pain (Psychiatric disorders) | 3 | 2
Hypotension (Vascular disorders) | 4 | 0
Constipation (Gastrointestinal disorders) | 1 | 4
Diarrhea (Gastrointestinal disorders) | 3 | 3
Melena (Gastrointestinal disorders) | 0 | 3
Nausea (Gastrointestinal disorders) | 7 | 3
Vomiting (Gastrointestinal disorders) | 6 | 2
Edema (Metabolism and nutrition disorders) | 3 | 0
Parasthesia (Nervous system disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less